CLINICAL TRIAL: NCT06180642
Title: Reliability and Validity of Ultrasound for the Assessment of Structural and Mechanical Properties of Soft Tissues at the Upper Limb Region in Women After Breast Cancer Treatment
Brief Title: Reliability and Validity of Ultrasound for the Assessment of Soft Tissue Properties After Breast Cancer Treatment
Acronym: SOFT-TI
Status: Recruiting | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, An De Groef, Professor, Universiteit Antwerpen
Other Study IDs: 2776
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms
Keywords: ultrasound; upper limb dysfunctions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women after breast cancer with UL dysfunctions
  Interventions: Other: Assessment of soft tissue properties; Other: Retest assessment of soft tissue properties
- Women after breast cancer without UL dysfunctions
  Interventions: Other: Assessment of soft tissue properties; Other: Retest assessment of soft tissue properties
- Healthy volunteers: age- and gender-matched control group
  Interventions: Other: Assessment of soft tissue properties; Other: Retest assessment of soft tissue properties

INTERVENTIONS:
Other: Assessment of soft tissue properties — Assessment of soft tissue properties at the upper limb region with clinical assessments and ultrasound
Other: Retest assessment of soft tissue properties — Retest Assessment of soft tissue properties at the upper limb region with clinical assessments and ultrasound

SUMMARY:
After 1 year, more than 50% experience upper limb (UL) complaints after treatment for breast cancer. These complaints are disabling and cause limitations in daily life and this leads to a decrease in the patient's quality of life. The cause of these UL complaints is complex and multifactorial. Due to breast cancer treatment, the structural (tissue composition and volume) and mechanical (tissue stiffness) properties of the soft tissue may change. These changes can occur in the muscle, skin and surrounding fascia and especially in the soft tissue around the breast and axilla where that treatment is localised.

Ultrasound with specific 'add-on' techniques can objectively assess these features and provide a picture of their role in UL function after breast cancer. The first aim in this study is to investigate the reliability and validity of conventional 2D ultrasound for 1) soft tissue composition and 2) soft tissue thickness at the level of the breast and upper limb. The reliability and validity of shear wave elastography, a specific complement to conventional 2D ultrasound, to assess tissue stiffness will also be examined.

ELIGIBILITY:
1. Breast cancer patients without upper limb dysfunctions (n=30) Inclusion Criteria

   * Patients with unilateral primary breast cancer
   * Surgery including, either: Mastectomy with axillary lymph node dissection or sentinel lymph node biopsy or breast conserving surgery with axillary lymph node dissection or sentinel lymph node biopsy
   * At least 3 months after surgery or radiotherapy in order to take into account wound healing
   * Comprehensive of the Dutch language
   * QuickDASH score <15/100

   Exclusion Criteria:
   * Bilateral surgery, widespread distance metastases, previous breast surgery
   * Diagnosis of neurological or rheumatological condition
   * upper limb dysfunctions caused by other reasons
2. Breast cancer patients with upper limb dysfunctions (n=30) Inclusion Criteria

   * Patients with unilateral primary breast cancer
   * Surgery including, either: Mastectomy with axillary lymph node dissection or sentinel lymph node biopsy or breast conserving surgery with axillary lymph node dissection or sentinel lymph node biopsy
   * At least 3 months after surgery or radiotherapy in order to take into account wound healing
   * Comprehensive of the Dutch language
   * QuickDASH score >15/100

   Exclusion Criteria:
   * Bilateral surgery, widespread distance metastases, previous breast surgery
   * Diagnosis of neurological or rheumatological condition
   * upper limb dysfunctions caused by other reasons
3. Healthy volunteers (n=30)

Inclusion criteria:

* Healthy women (QuickDASH <15) age-matched with a breast cancer patient from the main study
* Comprehensive of the Dutch language

Exclusion criteria:

* upper limb dysfunctions
* Diagnosis of neurological or rheumatological condition, diabetes

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with history of primary breast cancer
Study Population: Women with a history of primary breast cancer with and without upper limb dysfunctions and an age- and gender-matched healthy control group
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Reliability of soft tissue thickness (mm) | 1 week
  Intra- and inter-rater reliability of thickness (mm) of the skin, fat tissue, breast parenchyma, retromammary fat, and pectoralis major muscle measured with 2D ultrasound
Reliability of soft tissue composition | 1 week
  Intra- and inter-rater reliability of tissue composition (echo-intensity) measured with 2D ultrasound
Reliability of soft tissue elasticity (m/sec) | 1 week
  Intra- and inter-rater reliability of soft tissue elasticity (m/sec) of the pectoralis major muscle and breast measured with shear-wave elastography

SECONDARY OUTCOMES:
Validity of soft tissue elasticity | 1 week
  Soft tissue elasticity (m/sec) measured with the shear-wave elastography will be compared with the soft tissue index (N/m) measured with the MyotonPro, skin stiffness (N) measure with the SkinFibrometer, severity of tissue toxicity after radiotherapy (0-4) with the Late Radiation Morbidity Scoring Scheme (RTOG) and degree of myofascial adhesions (0-9) measured with the MAP-BC

CONTACTS AND LOCATIONS:
Locations (1):
- Universiteit Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No